CLINICAL TRIAL: NCT06960044
Title: Procalcitonin Aided Antimicrobial Therapy vs Standard of Care: a Randomized Prospective Clinical Trial
Brief Title: Procalcitonin Aided Antimicrobial Therapy vs Standard of Care
Acronym: PCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Collaborators: Thermo Fisher Scientific FS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ASO.MedI.24.02
Record Dates: First submitted 2025-04-24; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Lower Respiratory Tract Infection (LRTI)
Keywords: procalcitonin; procalcitonin-guided antibiotic management
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Interventional, randomized, two-arm with a 1:1 ratio study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Procalcitonin-guided antibiotic management (Experimental): Patients hospitalized in Internal Medicine, Geriatrics, Infectious Disease unit, Pneumology, Semi Intensive Care unit, ICU, Emergency Medicine with clinical and instrumental diagnosis of lower respiratory tract infection (LRTI), randomized in the experimental arm
  Interventions: Procedure: Procalcitonin-guided antibiotic management
- Standard of care (Active Comparator): Patients hospitalized in Internal Medicine, Geriatrics, Infectious Disease unit, Pneumology, Semi Intensive Care unit, ICU, Emergency Medicine with clinical and instrumental diagnosis of lower respiratory tract infection (LRTI), randomized in the control arm
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Procedure: Procalcitonin-guided antibiotic management — After the randomization, PCT plasma concentration will be dosed and repeated every 24 hours and antimicrobial treatment will be withdrawn as soon as the PCT value will decrease > 80% of peak value or will fall below 0.25 ng/mL. Patients with a normal baseline PCT value (below 0.25 ng/mL) will start the antimicrobial therapy, as clinically appropriate and PCT plasma concentration will be repeated every 24 hours, as indicated in the protocol. The antimicrobial agents will be managed according to the clinical and radiological evolution of the LRTI.
  Arms: Procalcitonin-guided antibiotic management
Procedure: Standard of care — Patients assigned to the control group will be treated according to the best standard of care and PCT will not be evaluated for the whole duration of the study.
  Arms: Standard of care

SUMMARY:
Antibiotic resistance is driven by overuse, especially for viral respiratory infections. Procalcitonin (PCT), a biomarker for bacterial infections, helps guide antibiotic therapy more precisely, reducing unnecessary use and improving outcomes. Studies, including large trials and economic models across several countries, show PCT-guided treatment lowers mortality, antibiotic exposure, therapy duration and related complications, potentially reducing hospital costs despite initial testing expenses.

DETAILED DESCRIPTION:
Antibiotic resistance (ABR) poses a significant threat to global health and is largely driven by the overuse of antibiotics, particularly for acute respiratory tract infections (ARTIs), which are mostly viral. Despite this, antibiotics are frequently prescribed, often for unnecessarily long durations due to the lack of reliable markers indicating illness resolution. This has led to an interest in using biomarkers like procalcitonin (PCT) to guide antibiotic therapy more accurately.

PCT is a precursor of the hormone calcitonin and increases significantly in the presence of bacterial infections, offering a promising tool for distinguishing bacterial from viral infections and for monitoring infection progression and response to treatment. It rises within hours of infection onset, peaks by day two, and decreases with recovery, making it useful for deciding when to start or stop antibiotics.

Clinical studies, including the large PRORATA randomized controlled trial, have demonstrated that PCT-guided antibiotic protocols are safe and effective in reducing antibiotic use without compromising patient outcomes. A Cochrane review further supported this, showing that PCT-guided therapy reduces mortality, antibiotic consumption, and antibiotic-related adverse effects in patients with ARTIs.

However, PCT testing has yet to be widely adopted in hospitals due to concerns about its cost-effectiveness and implementation challenges. To address these concerns, a series of health economic evaluations have been carried out: they assess the clinical and economic impact of PCT-guided therapy, particularly its role in reducing complications such as ABR and Clostridium difficile infections (CDI).

Findings consistently show that PCT-guided antibiotic therapy not only improves patient outcomes but also reduces direct healthcare costs when compared to standard care. Recent modeling incorporating RWE from a U.S. hospital further confirmed these benefits in real-world settings, strengthening the case for broader adoption of PCT in hospital-based antibiotic stewardship programs.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* clinical and instrumental diagnosis of LRTI consistent with bacterial origin and requiring antimicrobial treatment;
* patient hospitalized in Internal Medicine, Geriatrics, Infectious Disease unit, Pneumology, Semi Intensive Care unit, ICU, Emergency Medicine;
* informed consent provided by the patient.

Exclusion Criteria:

* age < 18 years;
* lack of informed consent;
* severe immunosuppression (other than related to corticosteroid use);
* concomitant diagnosis of other infections requiring long term antimicrobial therapy (i.e. endocarditis, osteomyelitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Duration of antimicrobial treatment | Periprocedural
  Measure of the antimicrobial treatment duration in days

SECONDARY OUTCOMES:
Length of hospital stay | Periprocedural
  Measure of the hospital stay in days
Sequential Organ Failure Assessment | At baseline and every 24 hours
  Assessment of clinical outcome with the SOFA Score, based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. Score ranges from 0 (best) to 24 (worst) points.
Quick Sequential Organ Failure Assessment | At baseline
  Assessment of clinical outcome with the qSOFA Score, a simplified version of the SOFA Score. Score ranges from 0 (best) to 3 (worst) points.
National Early Warning Score | At baseline and every 24 hours
  Assessment of clinical outcome with the NEWS Score, which identifies three alert levels with their specific clinical responses depending on the degree of criticality in relation to the final score derived (from 0 (code green) to 6 (code red)).
Incidence of Clostridium difficile infections (CDI) | Periprocedural
  Measure of the incidence of CDI with stool tests and GHD tests
Incidence of multi-drug resistance (MDR) infections | In the next 30 days after the baseline
  Measure of the incidence of MDR infections
Mortality | During the study, 4 weeks and 3 months from baseline
  Mortality evaluation
Costs | Periprocedural
  Evaluation of the costs associated with antibiotic therapy and hospitalization, relative to ABR per patient with LRTI and relative to CDI per patient with LRTI

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center, Alessandria, Piedmont, Italy